CLINICAL TRIAL: NCT06341296
Title: Phase II Study of Irinotecan Liposomes Combined With 5-FU/LV+ Bevacizumab in First-line Treatment of Metastatic Colorectal Cancer
Brief Title: Phase II Study of Irinotecan Liposomes in First-line Treatment of Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Dr., West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K07
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- irinotecan liposome injection combined with 5-FU/LV+ bevacizumab (Experimental): Patients will be treated with irinotecan liposome injection combined with 5-FU/LV+ bevacizumab. Treatment lasted 8 cycles.
  Interventions: Drug: Irinotecan Liposome; Drug: 5-FU; Drug: LV; Drug: Bevacizumab

INTERVENTIONS:
Drug: Irinotecan Liposome — 70 mg/m^2 , d1, 14 days per cycle, 8 cycles.
Drug: 5-FU — 5-FU 400mg/m^2, then 2400mg/m^2, continuous intravenous infusion for 46-48h, d1-2, 14 days per cycle, 8 cycles.
Drug: LV — 400mg/m^2, d1, 14 days per cycle, 8 cycles.
Drug: Bevacizumab — 5mg/kg, d1, 14 days per cycle, 8 cycles.

SUMMARY:
To evaluate the objective response rate, disease control rate, progression-free survival, overall survival, surgical conversion rate and safety of irinotecan liposome combined with 5-FU/LV+ bevacizumab regimen in first-line treatment of advanced metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
This is a Phase II clinical study to evaluate the efficacy and safety of the combination regimen of irinotecan liposome injection in the first-line treatment of metastatic colorectal cancer. Patients will receive liposomal injections of irinotecan 70mg/m^2 d1, bevacizumab 5mg/kg d1, LV 400mg/m^2 d1, 5-FU 400mg/m^2, then 2400mg/m^2, continuous intravenous infusion for 46-48h, d1-2. 86 eligible patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 18~85 years old.
* Histopathologically confirmed patient with an inoperable metastatic colorectal adenocarcinoma.
* RAS/BRAF v600e mutant or right half colon cancer is known.
* pMMR/MSS is known.
* The unresectable stage of metastatic disease has not received any systemic antitumor therapy.
* For subjects previously receiving neoadjuvant or adjuvant therapy, the date of first discovery of disease progression must be at least 6 months removed from the date of last administration of neoadjuvant or adjuvant therapy.
* ECOG 0~1, patients ≥75 years old need an ECOG score of 0
* The presence of at least 1 measurable lesion that can be evaluated according to the RECIST v1.1 criteria.
* Normal bone marrow and organ function: ① Neutrophils (ANC) ≥1.5×10^9/L, platelets (PLT) ≥100×10^9/L, hemoglobin (Hb) ≥80g/L, albumin (ALB) ≥30 g/L, white blood cells (WBC) ≥3.0×10^9/L, and no bleeding tendency; ② AST, ALT and alkaline phosphatase (ALP) were all ≤2.5× upper limit of normal range (ULN), and ≤5×ULN when liver metastases occurred; The total bilirubin level doesn't exceed the upper limit of the agency's normal range; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥40 ml/min (calculated according to Cockroft-Gault)
* Understand the situation of this study, patients and/or legal representatives voluntarily agree to participate in this study and sign informed consent form.

Exclusion Criteria:

* Known or suspected central nervous system metastasis.
* Received irinotecan/irinotecan liposomes/bevacizumab before enrollment.
* Had undergone surgery and other oncologic treatments within the first 4 weeks of enrollment.
* Previous treatment-related toxicity didn't return to NCI-CTCAE v5.0 I or below(except hair loss and peripheral neuropathy).
* The use of CYP3A, CYP2C8, and UGT1A1 inhibitors or inducers couldn't be discontinued or were not discontinued within 2 weeks prior to enrollment.
* Severe gastrointestinal dysfunction, gastrointestinal perforation, intraperitoneal abscess, and fistula.
* Intestinal obstruction, signs and symptoms of intestinal obstruction, or the stent has been previously implanted and the stent has not been removed before the screening period.
* Interstitial lung disease.
* Tendency of arterial embolism and massive bleeding within 6 months before enrollment (except surgical bleeding).
* Patients with fluid accumulation that couldn't reach a stable state but small amount of ascites on imaging without clinical symptoms could be enrolled.
* Any serious or uncontrolled systemic disease, including uncontrolled high blood pressure, heart disease, active bleeding, active viral infection, etc.
* Have had other malignancies within the past 5 years or currently, except cured cervical carcinoma in situ, uterine carcinoma in situ, and non-melanoma skin cancer.
* Patients of childbearing age who refuse to take contraceptives, women who are pregnant or breastfeeding.
* The researchers didn't consider it appropriate to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From initial medication to the date of first documented progression or end of medication or completed 8 cycles treatment, whichever came first . Assessed up to 4 months
  To investigate antitumor efficacy of study.

SECONDARY OUTCOMES:
Disease control rate | From initial medication to the date of first documented progression or end of medication or completed 8 cycles treatment, whichever came first. Assessed up to 4 months
  To investigate antitumor efficacy of study.
Progression free survival | From initial medication to the date of first documented progression or end of medication, whichever came first. Assessed up to 30 months.
  To investigate antitumor efficacy of study.
Overall survival | From initial medication to the date of death from any cause. Assessed up to 30 months.
  To investigate antitumor efficacy of study.
Percentage of patients undergoing surgery. | From the first dose to completed 8 cycles treatment. Assessed up to 5 months.
  To assess surgical conversion rates in patients who could be surgically resected.
R0 resection | From the first dose to the surgery. Assessed up to 6 months.
  To assess surgical conversion rates in patients who could be surgically resected.
Incidence of adverse events and severity of adverse events as assessed by CTCAE 5.0 | From the first dose to completed 8 cycles treatment. Assessed up to 5 months.
  To assess the incidence and severity of adverse events in combination regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Sichuan, Sichuan, Chengdu, China